CLINICAL TRIAL: NCT06848673
Title: PILOT CLINICAL TRIAL (PCT) of the Natural History of the Most Common MTBI-related Oculomotor Disorder Convergence Insufficiency & the Effectiveness of Vergence/Accommodative Therapy for MTBI-related Convergence Insufficiency
Brief Title: Natural History of MTBI-related Convergence Insufficiency & Effectiveness of Vision Therapy for MTBI-related CI
Acronym: TBEye
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR230111; VR230111 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Convergence Insufficiency
Keywords: Convergence Insufficiency; Vision Therapy; mTBI; Concussion; Office-based vergence/accommodative therapy
MeSH Terms: conditions — Ocular Motility Disorders; Brain Concussion | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomization to immediate OBVAM or delayed OBVAM
Who Masked: Investigator
Masking Description: The examiner who performs the sensory-motor vision examination will be masked to the assigned treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Office-Based Vergence/Accommodative Therapy with Movement (OBVAM) (Experimental): 16 sessions, twice per week of office-based vergence/accommodation therapy (OBVASM)While OBVAM therapy retains the essential elements of OBVAT. The OBVAM therapy protocol has four phases. Phase 1 targets visual/vestibular issues typical in mTBI-CI by integrating version eye movements, such as saccades and pursuits, with head and body movements. It also includes gross convergence, monocular accommodative (focusing) flexibility, and simple convergence procedures. The subsequent phases concentrate on enhancing ramp vergence amplitudes and improving accommodative facility (Phase 2), focusing on vergence facility and endurance (Phase 3), and integrating vergence and accommodation (Phase 4). Head and body movements are incorporated into some therapy procedures in Phases 3 and 4.
  Interventions: Other: Office-Based Vergence/Accommodative Therapy with Movement (OBVAM)
- Delayed Office-Based Vergence/Accommodative Therapy with Movement (OBVAM) (Active Comparator): Same as immediate group but delayed 6 weeks
  Interventions: Other: Office-Based Vergence/Accommodative Therapy with Movement (OBVAM)

INTERVENTIONS:
Other: Office-Based Vergence/Accommodative Therapy with Movement (OBVAM) — Head and body movements are incorporated into some therapy procedures in Phases 3 and 4. Additional details are provided in the Overall Program Narrative. Participants undergoing office-based VAM therapy will be prescribed home therapy procedures including the HTS2 Home Vision Therapy System (https://htsvision.com/) thrice weekly to support their in-office VAM therapy. This software progressively increases fusional convergence and divergence demands, offers instant user feedback, and will allow us to track participants' usage and progress. Basic procedures like free-space fusion cards and Brock String will also be prescribed for home therapy.

SUMMARY:
The design of this project is a pilot study, a type of feasibility study conducted in preparation for subsequent RCTs that will assess the effectiveness of office-based vergence/accommodative therapy with movement (OBVAM) for mTBI-related convergence insufficiency.

DETAILED DESCRIPTION:
The design of this project is a pilot study, a type of feasibility study conducted in preparation for subsequent RCTs that will assess the effectiveness of interventions or therapies. In this application, we refer to this pilot and feasibility study as a pilot clinical trial (PCT). This feasibility PCT aims to identify potential challenges, logistical issues, and unforeseen complications. To do this, we will examine various feasibility aspects, including recruitment and retention, randomization, intervention protocols, outcome measures, ethical considerations, safety monitoring, resource availability, and stakeholder feedback. By conducting this PCT, we can test our procedures and gather preliminary data. The primary objectives of this feasibility PCT are to 1) Determine the feasibility of conducting future full-scale RCTs by evaluating the effectiveness of a novel vergence/accommodative/move (OBVAM) therapy program for young adults with mTBI-CI and 2) Better understand the progression and stability (i.e., natural history) of mTBI-CI over the 6 weeks following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 35 years inclusive

  * Medical diagnosis of mTBI or concussion > 1 month ago and no longer than 6 months ago
  * Convergence Insufficiency Symptom (CISS score) ≥ 21
  * Best-corrected VA of 20/25 or better in both eyes at distance & near
  * Willingness to wear refractive correction, if indicated
  * Random dot stereopsis of 500 arcsec or better (Randot Stereo Test)
  * Receded NPC of ≥6 cm
  * Insufficient PFV (< 15∆ or PFV blur point less than twice the near exophoria magnitude)
  * Wearing refractive correction for cycloplegic refractive errors of:
  * ≥ +1.25 D SE hyperopia or ≥ -1.00 D SE myopia in either eye
  * ≥ 1.25 D astigmatism in either eye, ≥ 1.00 D SE anisometropia
  * Astigmatism axis within ±10 degrees if magnitude is ≤1.00 D and within ±5 degrees if >1.00 D

Exclusion Criteria:

* • No previous treatment for CI

  * No previous diagnosis of CI from an ophthalmologist or optometrist
  * No medications known to affect accommodation or vergence
  * Investigator & patient willing to forgo all other CI treatment other than that assigned by randomization

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Composite Measure | 6 weeks
  The primary outcome measure is a composite score of two key clinical measures: the near point of convergence (NPC) and positive fusional vergence at near (PFV). At the two outcome visits, each participant's performance on these clinical measures will be categorized according to the following predefined success criteria: 1) Successful: meets both criteria; a) NPC is <6 cm and improved ≥4 cm and b) PFV meets Sheard's criterion and the blur (break, if no blur) is >15Δ and increased ≥10Δ; 2) Improved: NPC improved ≥4 cm and PFV improved ≥10Δ; and 3) Non-Responder: Does not meet criteria for successful or improved

SECONDARY OUTCOMES:
Comparison of the Change in the Near Point of Convergence (NPC) break and recovery value | 6 weeks
  A standard near point rod will be used to measure the ability to converge the eyes. We will measure the NPC break (when double vision occurs) and the NPC recovery (when single vision is restored) . A comparison of the change in the break and recovery between the immediate and the delayed groups will be analyzed from baseline to to the first outcome visit (after 6 weeks).
Comparison of the Change in Positive Fusional Vergence after 6 weeks between the Two Groups | 6 weeks
  A hand-held prism bar will be used to assess positive fusional vergence (PFV) at baseline and after 6 weeks. We will measure the PFV break (when double vision occurs) and the PFV recovery (when single vision is restored) . A comparison of the change in the break and recovery between the immediate and the delayed groups will be analyzed from baseline to to the first outcome visit (after 6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, PhD, Principal Investigator — Drexel University

IPD SHARING:
Plan to Share IPD: No